CLINICAL TRIAL: NCT01991847
Title: Feasibility Study of the PROTECT-trial (The Potential and Role Of Tertiary Prevention by Exercise in Colorectal Cancer Therapy)
Brief Title: Tertiary Prevention by Exercise in Colorectal Cancer Therapy
Acronym: F-PROTECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Collaborators: German Cancer Aid (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: F-PROTECT
Record Dates: First submitted 2013-11-18; First posted 2013-11-25 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Colorectal Cancer
Keywords: colon; cancer; prevention; exercise; physical activity; rectal
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Physical activity (Experimental): Physical activity
  Interventions: Behavioral: Physical activity

INTERVENTIONS:
Behavioral: Physical activity — The patients will perform increasing volumes of moderate intensity endurance (e.g. walking, cycling) exercise, leading up to 18 MET-hours per week by the end of three months. Patients will then maintain this activity level for the remaining 9 months, with reduced supervision.

SUMMARY:
The purpose of this study is to determine the feasibility of a one year exercise training program in post-surgical patients with colorectal cancer.

DETAILED DESCRIPTION:
Apart from a genetic predisposition lifestyle factors (low physical activity, nutrition, and obesity) increase the risk of colorectal cancer. Furthermore, in observational studies increased physical activity has shown to improve the prognosis in patients after the diagnosis of colorectal cancer. However, there are currently no prospective randomized controlled trials which prove the causal relationship between exercise and prognosis in colorectal cancer patients. The long-term aim of this study is to evaluate whether physical activity of ≥ 18 MET-h (Metabolic equivalent task-hours) per week significantly improves disease free survival in colorectal cancer survivors (stage UICC II/III). In the first instance, structure-, process- as well as outcome-characteristics need to be investigated within a feasibility study (F-PROTECT). Essential aims are to establish collaborations with clinics and training centres, to achieve the required recruitment numbers, and to conduct the training intervention.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed nonhereditary primary Stage II or III colon cancer diagnosis or rectal cancer
* written informed consent in German
* histopathologically confirmed R0-resection
* start of guideline conformed adjuvant chemotherapy within 12 weeks after R0-resection in Stage III colon cancer diagnosis (if necessary in Stage III colon cancer diagnosis)

Exclusion Criteria:

* hereditary colon cancer diagnosis
* R1 and R2 resection
* clinically relevant complications during recovery
* secondary neoplasm
* non-continuance of guideline conformed therapy
* uncontrolled infection
* manifest cardiac disease (e.g. unstable CAD, heart failure (NYHA IV), malignant hypertension)
* clinical relevant respiratory disease (GOLD IV)
* musculoskeletal disorders severely restricting the patients mobility (e.g. gonarthrosis, coxarthrosis)
* cirrhosis of the liver (Child B and C)
* Karnofsky performance status scale ≤ 60%
* maximal exercise capacity ≤ 50 watt
* clinically relevant lab factors (leukocyte count ≤ 3000/μl, thrombocyte count ≤ 20.000/μl, hemoglobin < 8 g/dl)
* physical activity level ≥ 18 MET-h/ week at screening

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Target sample size | one year
  The primary outcome measure is to successfully recruit 50 colorectal cancer patients, and to achieve 70% compliance to regular exercise over one year.

SECONDARY OUTCOMES:
Physical activity | at screening and 3, 6, 9, and 12 month after baseline
  Physical activity will be measured using physical activity diary, heart rate monitor (Sigma Sport PC 22.13), accelerometer (Aipermotion 440), and the German version of the International Physical Activity Questionnaire (IPAQ).
Peak oxygen consumption | at baseline and 12 month after baseline
  Spiroergometry will be used to assess peak oxygen consumption (VO2peak).
Patient satisfaction | at 3, 6, 9, and 12 month after baseline
  Patient satisfaction will be measured using questionnaire.
Cancer related fatigue | at screening and 6 and 12 month after baseline
  Fatigue will be measured using the German version of the European Organization for Research on Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-FA13; reduced version with 13 items).
Anxiety and depression | at screening and 6 and 12 month after baseline
  Anxiety and depression will be assessed with the German version of the Hospital Anxiety and Depression Scale (HADS-D).
Cancer related quality of life | at screening and 6 and 12 month after baseline
  Cancer related quality of life will be assessed with the German Version of the European Organization for Research on Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ C30).
Quality of life in colorectal cancer | at screening and 6 and 12 month after baseline
  Cancer related quality of life will be assessed with the German Version of the European Organization for Research on Treatment of Cancer Quality of Life Questionnaire in colorectal cancer (EORTC QLQ-CR29).
Adverse and serious adverse events | one year
  Adverse (e.g. dizziness, high blood pressure) and serious adverse events (e.g. death, prolonged hospitalization) will be reported within 24 hours to the study physician via form.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Halle, Prof. M.D., Principal Investigator — Department of Prevention, Rehabilitation and Sports Medicine, Klinikum rechts der Isar, Technical University of Munich
Locations (1):
- Department of Medicine, Division of Prevention and Sports Medicine TU Munich, Munich, Germany

REFERENCES:
- [Derived] Heitkamp M, Spanier B, von Korn P, Knapp S, Gross C, Haller B, Halle M. Feasibility of a 12-Month Exercise Intervention in Postsurgical Colorectal Cancer Patients. Transl Sports Med. 2023 Jan 20;2023:4488334. doi: 10.1155/2023/4488334. eCollection 2023. PMID 38654917